CLINICAL TRIAL: NCT01872221
Title: Study of the Capacity of the MRI Spectroscopy to Define the Tumor Area Enriched in Glioblastoma Stem Cells. Proof of Concept Study
Acronym: STEMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12TETE01
Record Dates: First submitted 2013-05-07; First posted 2013-06-07 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Spectroscopy; MRI; Glioma stem cells; Surgery; Radioresistance
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery and radio-chemotherapy (Experimental): Surgery (on the basis of all preoperative multimodal MRI) followed by standard radio-chemotherapy stupp protocol
  Interventions: Procedure: Surgery (based on preoperative multimodal MRI) followed by the standard radio-chemotherapy stupp protocol

INTERVENTIONS:
Procedure: Surgery (based on preoperative multimodal MRI) followed by the standard radio-chemotherapy stupp protocol

SUMMARY:
This is a prospective biomedical study of interventional type which includes 16 patients on 52 months (24 months of inclusion and 28 months of follow up).

This pilot study, combining a metabolic imaging approach (Proton Magnetic Resonance Spectroscopy = 1HMRSI) and a biological one, will be performed in patients harbouring a Glioblastoma (GBM)to determine whether MRI markers of aggressiveness (CNI2) are associated with specific biological patterns as regards to GBMSC (GBM contains tumor stem cell).

In the first part of the study, patients with radiological criteria of GBM amenable to surgical resection will be included ; pre-operative multimodal MRI scans will be done and all data acquired (including H1MRS and DTI data) will be integrated in the image-guided surgical device (ie neuronavigation system) to be used intraoperatively. During tumor resection, tissue samples will be individualized, based on their multimodal imaging characteristics and sent to the radiobiology laboratory INSERM for biological analysis.

After surgery, patient will be treated by the standard radio-chemotherapy stupp protocol and will be followed according to standard practices; multimodal MRI will be performed every 2 months during the first year and then every 3 months until progression.

ELIGIBILITY:
Inclusion Criteria:

First part of the study (Surgery and Imagery):

1. Surgical indication for patients who present radiological criteria of glioblastoma.
2. Patient who are ≥18 years old
3. Patient must have performance status between 0 and 2 on the ECOG Performance Scale
4. Life expectancy ≥ 3 months
5. Patient affiliated to social security regimen
6. Patient has voluntarily agreed to participate by giving written informed consent for the first part of the study.

Second part of the study (Treatment and Biology):

1. Histologically confirmed glioblastoma
2. Patient must have performance status between 0 and 2 on the ECOG Performance Scale or 3 only is due to motor deficit.
3. Life expectancy ≥ 3 months
4. Patient affiliated to social security regimen
5. Patient has voluntarily agreed to participate by giving written informed consent for the second part of the study.

Exclusion Criteria:

First part of the study (Surgery and Imagery):

1. Patients who are not allowed to perform an MRI
2. Spectroscopic exam whose results are not contributive
3. Pregnant or nursing patient,
4. Patients under law protection
5. Patient who presents conditions that would interfere with cooperation with the requirements of the trial.
6. Patient who presents medical, severe or chronic biological or psychiatric conditions not allowing his enrolment in the study, according to the investigator's opinion

Second part of the study (Treatment and Biology):

1.Biological material received in the lab more than 48 hours after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Biologic analysis of the GBM resected samples for the capacity to form neurospheres in vitro | 4,5 years
  comparison CNI2 versus nCNI areas on the capacity to form neurospheres (yes or no) in vitro in stem cells medium up to 5 passages.
Biologic analysis of the GBM resected samples on the RNA expression of 5 stem cells markers | 4,5 years
  comparison CNI2 versus nCNI areas on the following criteria : scoring from 0 to 5 according to the RNA expression of 5 stem cells markers (CD133, Nestine, Sox2, Olig2 and Musashi)
Biologic analysis of the GBM resected samples for their capacity to form invasive brain tumor after orthotopic implantation of the cells in nude mice | 4,5 years

SECONDARY OUTCOMES:
Time to progression | 4,5 years
  The time to progression is defined as the time from surgery until progression
Overall survival | 4,5 years
  The overall survival is defined as the time from surgery until death from any cause or last of follow-up news (censored data)

OTHER OUTCOMES:
Ancillary study of neurocognitive function | 4,5 years
  The neurocognitive function will be evaluated using the following tests:
  * trail making test
  * stroop color test
  * line-bissection task
  * Subtests of the WAISIII
  * MT 86 (Joanette 1992)
  * HDAE (BDAE) (Goodglass 1972)
  * MEC (Joanette 2004)
  * ECOSSE (Lecocq 1996) Quality of life will be evaluated using EORTC questionnaire QLQ C-30 and QLQ BN20.
Ancillary study of quality of life | 4,5 years
  Quality of life will be evaluated using EORTC questionnaire QLQ C-30 and QLQ BN20

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth MOYAL, professor, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - CHU Rangueil, Toulouse
  - Institut Claudius REGAUD, Toulouse

REFERENCES:
- [Derived] Pinto G, Saenz-de-Santa-Maria I, Chastagner P, Perthame E, Delmas C, Toulas C, Moyal-Jonathan-Cohen E, Brou C, Zurzolo C. Patient-derived glioblastoma stem cells transfer mitochondria through tunneling nanotubes in tumor organoids. Biochem J. 2021 Jan 15;478(1):21-39. doi: 10.1042/BCJ20200710. PMID 33245115